CLINICAL TRIAL: NCT06713135
Title: An Open-label Study to Collect Safety and Effectiveness Information on Long-term Treatment With Vamorolone in Boys With Duchenne Muscular Dystrophy Who Have Completed Prior Studies With Vamorolone
Brief Title: A Study on Safety and Effectiveness of Long-term Treatment With Vamorolone in Boys With Duchenne Muscular Dystrophy
Acronym: GUARDIAN
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNT-IV-VAM-011
Record Dates: First submitted 2024-11-16; First posted 2024-12-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne; vamorolone; santhera; long-term safety
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — VBP15 compound; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- vamorolone (Experimental): On Day 1, Subjects will roll over from a previous vamorolone program and continue treatment with vamorolone under this protocol. During the study, vamorolone will be administered at a dose range between 2 mg/kg/day and 6 mg/kg/day for boys weighing <40 kg. For boys weighing 40 kg or above, the dose range will be 80 mg to 240 mg once daily.
  Interventions: Drug: vamorolone 40 mg/mL oral suspension

INTERVENTIONS:
Drug: vamorolone 40 mg/mL oral suspension — Vamorolone is administered at a dose range between 2 mg/kg/day and 6 mg/kg/day for boys weighing <40 kg. For boys weighing 40 kg or above, the dose range will be 80 mg to 240 mg once daily. Doses can be adjusted within the dose range as determined by the Investigator based on tolerability. The highest tolerated dose should be used.
  Other Names: vamorolone

SUMMARY:
This study aims to assess safety and effectivness of long-term treatment with vamorolone in boys with Duchenne Muscular Dystrophy (DMD) who have completed prior studies with vamorolone.

DETAILED DESCRIPTION:
All subjects in this study have completed previous studies with vamorolone and continued to receive vamorolone under special programs: Compassionate Use Program [CUP], Named Patient Program [NPP] or Expanded Access Protocol [EAP]. All subjects will continue treatment with vamorolone under Guardian protocol instead. The primary objective of this study is to evaluate the safety of long-term treatment with vamorolone in boys with Duchenne Muscular Dystrophy regarding vertebral fractures. Secondary study objectives will evaluate the safety of long-term treatment with vamorolone on non-vertebral fractures, cataracts, delayed puberty, overall safety as well as ambulatory and non-ambulatory function.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or subject's parent(s) or legal guardian has provided written informed consent
* Subject has previously completed either the VBP15-LTE or VBP15-004 study, and transitioned through the Compassionate Use Program, Named Patient Program or Expanded Acess Protocol
* Subject is on vamorolone on day of enrolment
* Subject and parent / legal guardian are willing and able to comply with the protocol schedule, assessments and requirements

Exclusion Criteria:

* Any medical condition, which in the opinion of the Investigator, would affect study participation, performance or interpretation of study assessments
* Vamorolone treatment discontinued for ≥ 6 months within the year prior to enrolment for a non-safety reason, or vamorolone treatment previously discontinued at any time for a safety reason
* Severe hepatic impairment

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of vertebral fractures per 1000 person-years based on X-ray central reading. | At Enrolment and every 2 years during a Full visit
  Lateral thoracolumbar spine X-Rays will be collected and sent to a central reader for evaluation of vertebral fractures

SECONDARY OUTCOMES:
Time to first vertebral fractures (cumulative incidence) | From enrolment up to at least 2 years
Number of non-vertebral fractures per 1000 person-years based on investigator reporting | From enrolment until up to at least 3 years
  Non-vertebral fractures will be reported by investigators and not reviewed centrally
Time to first non-vertebral fractures (cumulative incidence) | From enrolment until up to at least 3 years
Number of cataracts per 1000 person-years based on ophthalmologist assessment | From enrolment until up to at least 3 years
  An ophthalmologist assessment including assessment of posterior capsular cataracts by slit lamp will be performed yearly
Number of subjects not reaching Tanner stage 2 by 15 years of age | From enrolment until up to at least 3 years
  Qualified personnel (eg, an individual, part of the endocrinology team and trained to assess Tanner stages) will provide an assessment of the puberty status of the subject, including testicular volume.
Frequency of adverse events (AEs) and serious adverse events (SAEs) | From enrolment until up to at least 3 years
  The occurrence of AEs should be sought by questioning of the subject and/or his caregiver at each visit or phone call during the study. All SAEs occurring from signature of the ICF up to 30 days after last dose of study medication must be reported, irrespective of severity or whether or not considered related to study medication. All SAEs must be reported within 24 hours of becoming aware of the event, whether or not the SAE is considered to be related to the study medication.
Change from baseline in body weight | From enrolment until up to at least 3 years
  Physical examination will include weight (in kg)
Number of subjects with clinically relevant laboratory abnormalities | From enrolment until up to at least 3 years
  Clinically relevant laboratory abnormalities will include HbA1c and morning cortisol measurements.
Change from baseline in Time to Stand (TTSTAND) velocity | From enrolment until up to at least 3 years
  The TTSTAND measures the time (in seconds) required for the subject to stand to an erect position from a supine position (floor)
Six-minute Walk Test (6MWT) | From enrolment until up to at least 3 years
  6MWT will be performed only in the ambulatory subjects. The total distance traveled, in meters, should be recorded along with the validity of the test as assessed by the test administrator. If a subject cannot complete 6 minutes of walking, the total meters and the time until discontinuation of the test should be recorded.
Change from baseline in 6MWT distance | From enrolment until up to at least 3 years
Age at ambulatory and non-ambulatory milestones | From enrolment until up to at least 3 years
  Ambulatory milestones include Loss of standing from the floor, Loss of ability to climb 4-stairs, Loss of ability to walk 10 meters (loss of ambulation), Loss of ability to stand unassisted. Non-ambulatory milestones include Loss of ability to perform hand-to-mouth function, Loss of ability to use a manual wheelchair, Loss of ability to transfer independently from wheelchair, Nocturnal ventilation and Full time ventilation.
North Star Ambulatory Assessment (NSAA) scores | At enrolment and each Full visit (Month 12, 24, 36, etc / End-of -Treatment) until End of Study
  The NSAA is a 17-item rating scale that is used to measure functional motor abilities in ambulant children with DMD and allows to monitor the progression of the disease and treatment effects.
Change from baseline in body height | From enrolment until up to at least 3 years
  Physical examination will include height (in cm). Ulnar length of the non-dominant arm will be used if standing height cannot be measured.
Change from baseline in Body Mass Index (BMI) | From enrolment until up to at least 3 years
  BMI will be derived based on weight and height at every study visit

CONTACTS AND LOCATIONS:
Overall Officials: A Child, MD, Principal Investigator — Leeds Teaching Hospital
Locations (18):
- Belgium (2):
  - UZ Gent (Universitair Ziekenhuis Gent), Ghent
  - UZ Leuven (Universitair Ziekenhuis Leuven), Leuven
- Czechia (2):
  - University Hospital Brno, Brno
  - Fakultni Nemocnice Motol, Prague
- Children's Hospital Agia Sofia, Athens, Greece
- Children's Health Ireland at Tallaght, Tallaght University Hospital, Dublin, Ireland
- Schneider Children's Medical Center, Petah Tikva, Israel
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Radboud University Nijmegen, Nijmegen
- Te Wao Nui - Child Health Service, Wellington Hospital, Wellington, New Zealand
- Spain (2):
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario y Politecnico de La Fe, Valencia
- United Kingdom (6):
  - Queen Elizabeth University Hospital, Glasgow, Lanarkshire
  - Alder Hey Children's Hospital, Liverpool, Merseyside
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - The John Walton Muscular Dystrophy Research Centre, Newcastle

REFERENCES:
- [Background] Guglieri M, Clemens PR, Perlman SJ, Smith EC, Horrocks I, Finkel RS, Mah JK, Deconinck N, Goemans N, Haberlova J, Straub V, Mengle-Gaw LJ, Schwartz BD, Harper AD, Shieh PB, De Waele L, Castro D, Yang ML, Ryan MM, McDonald CM, Tulinius M, Webster R, McMillan HJ, Kuntz NL, Rao VK, Baranello G, Spinty S, Childs AM, Sbrocchi AM, Selby KA, Monduy M, Nevo Y, Vilchez-Padilla JJ, Nascimento-Osorio A, Niks EH, de Groot IJM, Katsalouli M, James MK, van den Anker J, Damsker JM, Ahmet A, Ward LM, Jaros M, Shale P, Dang UJ, Hoffman EP. Efficacy and Safety of Vamorolone vs Placebo and Prednisone Among Boys With Duchenne Muscular Dystrophy: A Randomized Clinical Trial. JAMA Neurol. 2022 Oct 1;79(10):1005-1014. doi: 10.1001/jamaneurol.2022.2480. PMID 36036925
- [Background] Dang UJ, Damsker JM, Guglieri M, Clemens PR, Perlman SJ, Smith EC, Horrocks I, Finkel RS, Mah JK, Deconinck N, Goemans NM, Haberlova J, Straub V, Mengle-Gaw L, Schwartz BD, Harper A, Shieh PB, De Waele L, Castro D, Yang ML, Ryan MM, McDonald CM, Tulinius M, Webster RI, Mcmillan HJ, Kuntz N, Rao VK, Baranello G, Spinty S, Childs AM, Sbrocchi AM, Selby KA, Monduy M, Nevo Y, Vilchez JJ, Nascimento-Osorio A, Niks EH, De Groot IJM, Katsalouli M, Van Den Anker JN, Ward LM, Leinonen M, D'Alessandro AL, Hoffman EP. Efficacy and Safety of Vamorolone Over 48 Weeks in Boys With Duchenne Muscular Dystrophy: A Randomized Controlled Trial. Neurology. 2024 Mar 12;102(5):e208112. doi: 10.1212/WNL.0000000000208112. Epub 2024 Feb 9. PMID 38335499
- [Background] Hoffman EP, Schwartz BD, Mengle-Gaw LJ, Smith EC, Castro D, Mah JK, McDonald CM, Kuntz NL, Finkel RS, Guglieri M, Bushby K, Tulinius M, Nevo Y, Ryan MM, Webster R, Smith AL, Morgenroth LP, Arrieta A, Shimony M, Siener C, Jaros M, Shale P, McCall JM, Nagaraju K, van den Anker J, Conklin LS, Cnaan A, Gordish-Dressman H, Damsker JM, Clemens PR; Cooperative International Neuromuscular Research Group. Vamorolone trial in Duchenne muscular dystrophy shows dose-related improvement of muscle function. Neurology. 2019 Sep 24;93(13):e1312-e1323. doi: 10.1212/WNL.0000000000008168. Epub 2019 Aug 26. PMID 31451516
- [Background] Mah JK, Clemens PR, Guglieri M, Smith EC, Finkel RS, Tulinius M, Nevo Y, Ryan MM, Webster R, Castro D, Kuntz NL, McDonald CM, Damsker JM, Schwartz BD, Mengle-Gaw LJ, Jackowski S, Stimpson G, Ridout DA, Ayyar-Gupta V, Baranello G, Manzur AY, Muntoni F, Gordish-Dressman H, Leinonen M, Ward LM, Hoffman EP, Dang UJ; NorthStar UK Network and CINRG DNHS Investigators. Efficacy and Safety of Vamorolone in Duchenne Muscular Dystrophy: A 30-Month Nonrandomized Controlled Open-Label Extension Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2144178. doi: 10.1001/jamanetworkopen.2021.44178. PMID 35076703
- [Background] Conklin LS, Damsker JM, Hoffman EP, Jusko WJ, Mavroudis PD, Schwartz BD, Mengle-Gaw LJ, Smith EC, Mah JK, Guglieri M, Nevo Y, Kuntz N, McDonald CM, Tulinius M, Ryan MM, Webster R, Castro D, Finkel RS, Smith AL, Morgenroth LP, Arrieta A, Shimony M, Jaros M, Shale P, McCall JM, Hathout Y, Nagaraju K, van den Anker J, Ward LM, Ahmet A, Cornish MR, Clemens PR. Phase IIa trial in Duchenne muscular dystrophy shows vamorolone is a first-in-class dissociative steroidal anti-inflammatory drug. Pharmacol Res. 2018 Oct;136:140-150. doi: 10.1016/j.phrs.2018.09.007. Epub 2018 Sep 13. PMID 30219580
- [Result] K. Nip, A. de Vera, S. Hasham, P. Charef, S. Wong. An open-label study to collect long-term safety and efficacy data from boys with DMD who have completed prior studies with vamorolone (GUARDIAN Study). Neuromuscular Disorders Volume 43, Supplement 1, October 2024, 104441.298